CLINICAL TRIAL: NCT05347342
Title: A Novel Multiplex Immunoassay for the Early Detection of Bladder Cancer
Brief Title: A Diagnostic for the Early Detection of Bladder Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Nonagen Bioscience Corporation (Industry); National Cancer Institute (NCI) (NIH); VA Long Beach Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Charles Rosser, Professor, Cedars-Sinai Medical Center
Other Study IDs: IIT2021-19-Furyua-EarlyDx; R01CA277810 (NIH)
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine collection (minimal 50 mL) yearly for 4 years of screening.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To improve upon the non-invasive detection of bladder cancer by further validating a multiplex ELISA assay directed at a bladder cancer-associated diagnostic signature in voided urine samples of patients with a high risk of developing bladder cancer.

DETAILED DESCRIPTION:
Environmental exposures, specifically tobacco smoke, increases the risk of many cancers, including bladder cancer. To date, there are no diagnostics capable of detecting bladder cancer early, that is prior to clinical presentation. Because of this severe limitation, nearly 30% of patients initially present with stage 2 and higher bladder cancer. Stage 2 bladder cancer has a 5-year survival of 50%, while stage 3/4 have a 5-year survival of <20%. Ideally, bladder cancer would be preventable. Unfortunate, this has not come to fruition. If these stage 2-4 bladder cancer cases could be detected at Stage 1 (5-yr survival >94%), then its possible to see an improvement in bladder cancer survival rates (21-23).

in this study, a urine-based diagnostic that possesses the potential to accurately identify patients who harbor bladder cancer prior to clinical manifestation will be tested.

ELIGIBILITY:
Inclusion Criteria:

Participants must be:

1. Age 50 years or older
2. >20 pack year history of tobacco exposure
3. Free of any malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years. Patients with localized prostate cancer who are being followed by an active surveillance program are also eligible.
4. Scheduled to be evaluated in the Pulmonary Rehab Clinic or Lung Cancer Screening Clinic
5. Willing and able to give written informed consent
6. Willing to provide voided urine sample
7. Be able and willing to complete semi-annual research clinic visits for 4 years

Exclusion Criteria:

Participants must not have:

1. History of hematuria (microscopic or gross) within 2 years of signing consent.
2. Previous history of bladder cancer
3. A known active urinary tract infection or urinary retention
4. An active stone disease (renal or bladder) or renal insufficiency (creatinine >2.0 mg/dL) - Serum creatinine value can be up to 2 years before consent, otherwise repeat.
5. An ureteral stents, nephrostomy tubes or bowel interposition
6. A recent genitourinary instrumentation (within 7 days prior to collection of voided urine sample)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women 50 years and older who have greater than a 20 pack year history of tobacco use.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
1. To assess the ability to recruit and retain an appropriate high-risk group of subjects into a 4-year longitudinal study monitoring them for the development of bladder cancer. | 5 years
  Ability to recruit
2. To report the sensitivity and specificity of the multiplex immunoassay ability to detect bladder cancer in patients with high risk of developing bladder cancer: >50 years and >40 pack year history of tobacco exposure. | 5 years
  Performance of multiplex test in this study
3. To develop a prediction risk calculator from this cohort using cutting edge machine learning techniques (e.g., random forest) incorporating biomarker data and clinical data. | 5 years
  Development of a risk calculator

CONTACTS AND LOCATIONS:
Overall Officials: Hideki Furuya, Principal Investigator — Cedars-Sinai Medical Center
Locations (2):
- United States (2):
  - Long Beach VA Healthcare System, Long Beach, California
  - Cedars-Sinai Medical Center, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2025-12-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT05347342/ICF_000.pdf